CLINICAL TRIAL: NCT03893019
Title: Multicenter Phase I Trial of MB-CART20.1 for the Treatment of Patients With Metastatic Melanoma
Brief Title: MB-CART20.1 Melanoma
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The risk-benefit assessment was not as expected.
Sponsor: Miltenyi Biomedicine GmbH (Industry)
Collaborators: DLR German Aerospace Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M-2015-307
Record Dates: First submitted 2019-03-06; First posted 2019-03-27 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Melanoma (Skin)
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose Level 1: 1x10e5 MB-CART20.1 cells (Experimental): 3+3 patients will be treated with 1x10e5 MB-CART20.1 cells per kg body weight administered intravenously
  Interventions: Biological: MB-CART20.1
- Dose Level 2: 1x10e6 MB-CART20.1 cells (Experimental): 3+3 patients will be treated with 1x10e6 MB-CART20.1 cells per kg body weight administered intravenously
  Interventions: Biological: MB-CART20.1
- Dose Level 3: 1x10e7 MB-CART20.1 cells (Experimental): 3+3 patients will be treated with 1x10e7 MB-CART20.1 cells per kg body weight administered intravenously
  Interventions: Biological: MB-CART20.1

INTERVENTIONS:
Biological: MB-CART20.1 — MB-CART20.1 consists of autologous CD20 Chimeric Antigen Receptor (CAR) transduced CD4/CD8 enriched T cells targeting CD20.positive tumor cells
  Other Names: CD20-targeting CAR T cells; anti-CD20 CAR T cells

SUMMARY:
This is a phase l multi-centric, single arm, prospective, open, dose-escalation study in patients with unresectable stage III oder IV melanoma. The trial will include 15 adult patients. The trial is a classic 3+3 design with 1 Log dose increments and maximum 3 dose levels of the intravenously administered MB-CART20.1.

DETAILED DESCRIPTION:
This Phase I trial will be the first trial with CD20 CAR transduced T cells in Europe targeting melanoma. The rationale for the trial is based on the finding that melanoma cancer sustaining cells express CD20 and that targeting CD20+ cells in preclinical model has a strong antitumor effect.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients with

* Histologically confirmed unresectable stage III or stage IV melanoma
* Willingness to provide a tumor biopsy between the screening visit and prior to administration of the IMP and eight weeks after treatment
* Progressive disease despite treatment with indicated standard therapies. Time window for decision about progressive disease is to be made depending on the treatment regimen chosen.
* Measurable lesions according to RECIST1.1
* ECOG (Eastern cooperative oncology group) performance status of 0-2
* Negative serological hepatitis B (HBV) test defined as negative tests for HBsAg and HBcAb, unless serology is positive due to recent IVIG therapy, HBcAb positivity will be allowed if HbsAb is present, negative testing of HCVAb, negative human immunodeficiency virus (HIV) 1/2 test within 6 weeks prior to enrollment.
* Estimated life expectancy of more than 6 months
* At least 18 years of age
* WBC ≥ 2500/µL
* ANC ≥ 1000/µL
* Platelets ≥ 75 x 103/µL
* Hemoglobin ≥ 9 g/dL
* AST ≤ 3 x upper limit of normal (ULN) for patients without liver metastasis
* AST < 5 x ULN for patients with liver metastasis
* Total Bilirubin ≤ 2 x ULN
* patients with Gilbert's Syndrome increase of indirect bilirubin < 6mg/dL
* No childbearing potential (i.e. postmenopausal, absence of menstrual bleeding for at least 1 year, hysterectomy, bilateral ovariectomy or tubal section/ligation) or negative pregnancy test at screening and before chemotherapy in women with childbearing potential. Sexually active female patients of childbearing potential should use one of the following highly effective methods of contraception (Pearl index < 1%): hormonal contraceptives (oral, injected, implanted, transdermal), intrauterine devices or systems (e.g. hormonal and non-hormonal IUD), or vasectomized sexual partner for at least 1 month before the trial start, during the course of the trial and in the 6 months following dosing. Sexual abstinence is restricted to true abstinence ( in line with the preferred and usual lifestyle of the subject).
* male patients, unless surgically sterile, must be using two acceptable methods for contraception (e.g. spermicide and condom) during the trial and refrain from fathering a child throughout the trial and for up to 12 months after dosing.
* Signed and dated informed consent before conduct of any trial-specific procedure.

Exclusion Criteria:

* Any evidence of brain metastases
* CNS (central nervous system) disorders and previous strokes, if clinically relevant
* Patients with epilepsy
* Clinically relevant autoimmune disorders or history of clinically relevant autoimmune disorders
* Patients with T-cell lymphoma
* Treatment with anti-CD20 antibodies or checkpoint blockade inhibitors within 6 weeks before leukapheresis
* Chemotherapy within 6 weeks prior to leukapheresis
* History of primary immunodeficiency
* Creatinine clearance < 50 ml/min calculated according to the modified formula of Cockcroft and Gault
* concurrent systemic radiotherapy
* Use of systemic corticosteroids and immunosuppressive medication except prednisone ≤ 10 mg QD or equivalent
* Patients with severe cardiac disease (e.g. NYHA Functional Class III or IV, myocardial infarction within 6 months before inclusion, ventricular tachyarrhythmia requiring ongoing treatment, unstable angina pectoris)
* Other investigational treatment within 4 weeks before MB-CART20.1 infusion
* Hypersensitivity against any drug or its ingredients/impurities that is scheduled or likely to be given during trial participation, e.g. as part of the mandatory lymphodepletion protocol, pre-medication for infusion, rescue medication/salvage therapies for treatment related toxicities
* Patients in which such medication (likely to be given during trial participation) is contraindicated for other reasons than hypersensitivity, e.g. live vaccines and fludarabine.
* Severe pulmonary disease (DLCO and/or FEV1 < 65%, dyspnoea at rest)
* Active systemic fungal, viral or bacterial infection
* Pregnant or lactating women
* Patient's lack of accountability, inability to appreciate the nature, meaning and consequence of the trial and to formulate his/her own wishes correspondingly
* Patients who have a relationship of dependence or employer employee relationship to the sponsor or the investigator
* Committal to an institution on judicial or official order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Determination of MTD | Week 4 after infusion of MB-CART20.1
  MTD is defined as the highest dose level at which < 33% of patients experience dose limiting toxicity (DLT)
Safety and Toxicity Assessment per Adverse Event reporting classified according to CTCAE V5.0 | until day 28 after infusion of MB-CART20.1
  per Adverse Event reporting classified according to CTCAE V5.0

SECONDARY OUTCOMES:
Clinical Response | 1 year after infusion of MB-CART20.1
  Number of patients with either Complete Response, Partial Response, Stable Disease or Progressive Disease using RECIST 1.1
Frequency of B-cell aplasia | 1 year after infusion of MB-CART20.1
  Circulating B cell numbers in the peripheral blood will be assessed by Flow cytometry
Phenotype and Persistence of infused MB-CART20.1 | 1 year after infusion of MB-CART20.1
  Blood samples for determination of persistence/phenotyping of infused MB-CART20.1 will be analysed.
Presence and phenotype of MB-CART20.1 and B cells in biopsies | Screening, 8 weeks after infusion of MB-CART20.1
  Tumor biopsies for determination of persistence/phenotyping of infused MB-CART20.1 will be analysed
Number of CD20+ tumor cells | Screening, 8 weeks after infusion of MB-CART20.1
  Tumor biopsies for determination of number of CD20+ tumor cells
Persistence of T-cell expansion for each dose group | Day 0 and week 12
  Blood samples for determination MB-CART20.1 levels (transgene copies / genomic DNA)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Borchmann, Prof., Principal Investigator — Universitätsklinikum Köln
Locations (1):
- University Hospital of Cologne - Clinic for Internal Medicine I, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aleksandrova K, Leise J, Priesner C, Aktas M, Apel M, Assenmacher M, Burger I, Richter A, Altefrohne P, Schubert C, Holzinger A, Barden M, Bezler V, von Bergwelt-Baildon M, Borchmann P, Goudeva L, Glienke W, Arseniev L, Esser R, Abken H, Koehl U. Automated manufacturing and characterization of clinical grade autologous CD20 CAR T cells for the treatment of patients with stage III/IV melanoma. Front Immunol. 2024 Sep 25;15:1328368. doi: 10.3389/fimmu.2024.1328368. eCollection 2024. PMID 39386211